CLINICAL TRIAL: NCT01574235
Title: Safety of Nivestim® in Patients Treated With Neutropenia-inducing Anticancer Chemotherapy in Routine Practice
Brief Title: Nivestim® (Filgrastim) Tolerance in Patients Treated by Toxic Chemotherapeutic Agents
Status: Completed | Type: Observational
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: NEXT
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Solid Tumors; Malignant Hemopathy; Chemotherapy-induced Febrile Neutropenia (FN)
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Curative or prophylactic Nivestim® treatment for FN
  Interventions: Biological: Nivestim®

INTERVENTIONS:
Biological: Nivestim®

SUMMARY:
The main aim of the study is to assess the safety of Nivestim® treatment in patients treated with neutropenia-inducing chemotherapy for a malignant disease, solid tumor or a malignant hemopathy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients presenting with a solid tumor or a malignant hemopathy,
* Patients treated with or beginning treatment with neutropenia-inducing chemotherapy (regardless of the cycle),
* Patients in whom treatment with Nivestim® is instituted for the purpose of reducing the duration of the neutropenias and the incidence of the chemotherapy-induced febrile neutropenias

Exclusion Criteria:

* Patients presenting with a chronic myeloproliferative syndrome,
* Patients presenting with a myelodysplastic syndrome,
* Patients showing hypersensitivity to any of the ingredients of Nivestim®,
* Patients not receiving chemotherapy,
* Patients who were already included in the study during a previous chemotherapy line

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving chemotherapy and treated with Nivestim® to prevent or reduce chemotherapy-induced febrile neutropenia.
Sampling Method: Non-Probability Sample
Enrollment: 2114 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety of Nivestim® to reduce or prevent febrile neutropenia in patients treated with neutropenia-inducing chemotherapy for a malignant disease, solid tumor or a malignant hemopathy. | Each patient will be followed for the duration of his chemotherapy regimen (the current one at the time of the Nivestim® treatment initiation) up to a maximum of six months
  The safety will be assessed by the record of all treatment emergent adverse events and all data about hospitalization due to any febrile neutropenia or infection.

SECONDARY OUTCOMES:
Efficacy of treatment with Nivestim® | Each patient will be followed for the duration of his chemotherapy regimen (the current one at the time of the Nivestim® treatment initiation) up to a maximum of six months
  Assess the efficacy of the treatment with Nivestim® by studying occurrence of febrile neutropenia, infection and the impact of these events on the chemotherapy treatment (cycle postponement, dose reduction)
Characteristics of the patients treated with Nivestim® in real-life practice | At Visit 1
  Describe the characteristics of the patients treated with Nivestim® in real-life practice,
Methods of treatment with Nivestim® | Each patient will be followed for the duration of his chemotherapy regimen (the current one at the time of the Nivestim® treatment initiation) up to a maximum of six months
  Describe the methods of treatment with Nivestim® depending on the indications (curative or prophylactic) in routine practice.
Profiles of the physicians participating in the study | At visit 1
  Describe the profiles of the physicians participating in the study
General practice of these physicians with regard to prescription of Granulocyte-Colony Stimulating Factors (G-CSF) | At visit 1
  Assess the general practice of these physicians with regard to prescription of G-CSF

CONTACTS AND LOCATIONS:
Locations (87):
- France (87):
  - Hopital Louis Pasteur, Colmar, Alsace
  - Hopital Jean Monnet, Épinal, Alsace
  - CH Emile Muller, Mulhouse, Alsace
  - CAC Paul Strauss, Strasbourg, Alsace
  - Chu Hopital Civil, Strasbourg, Alsace
  - STE ANNE, Strasbourg, Alsace
  - MEDIPOLE, Aix-les-Bains, Auvergne-Rhône-Alpes
  - CHRA, Annecy, Auvergne-Rhône-Alpes
  - Clinique CONVERT, Bourg-en-Bresse, Auvergne-Rhône-Alpes
  - Ch Chambery, Chambéry, Auvergne-Rhône-Alpes
  - Chu Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Ch Valence, Valence, Auvergne-Rhône-Alpes
  - Polyclinique Cesson, Cesson, Basse Normandie
  - Chu Rennes, Rennes, Basse Normandie
  - CHU SUD, Rennes, Basse Normandie
  - Clinique St Laurent, Rennes, Basse Normandie
  - Chp St Greg, Saint-Grégoire, Basse Normandie
  - Ch St Malo, St-Malo, Basse Normandie
  - CHG William MOREY, Chalon S/s, Bourgogne-Franche-Comté
  - CHU du BOCAGE, Dijon, Bourgogne-Franche-Comté
  - Clinique St Faron, Meaux, Champagne
  - Cac Jean Godinot, Reims, Champagne
  - Hopital St Quentin, Saint-Quentin, Champagne
  - Hopital Troyes, Troyes, Champagne
  - CHG Dieppe, Dieppe, Haute Normandie
  - Clinique Pasteur, Évreux, Haute Normandie
  - CH Jacques Monod, Montivilliers, Haute Normandie
  - Centre frederic joliot curie, Rouen, Haute Normandie
  - CHG, Alès, Languedoc
  - CHG, Béziers, Languedoc
  - CHG, Carcassonne, Languedoc
  - Chu St Eloi, Montpellier, Languedoc
  - Clinique Beausoleil, Montpellier, Languedoc
  - CHU Caremeau, Nîmes, Languedoc
  - Chg St Jean, Perpignan, Languedoc
  - Ch Du Pays D'Aix, Aix-en-Provence, Marseille
  - Clinique Rambot, Aix-en-Provence, Marseille
  - Ch Duffaut, Avignon, Marseille
  - Chp Clairval, Marseille, Marseille
  - Chu Timone, Marseille, Marseille
  - Fondation Saint Joseph, Marseille, Marseille
  - Hopital A.Pare, Marseille, Marseille
  - IPC, Marseille, Marseille
  - Chr Brive, Brivé, Massif Central
  - Chu Estaing, Clermont, Massif Central
  - Chu Gabriel Montpied, Clermont, Massif Central
  - Pole Sante Republique, Clermont, Massif Central
  - Clinique Vitalia Desertines, Montluçon, Massif Central
  - CHR, Roanne, Massif Central
  - Icl St Etienne, Saint-Etienne, Massif Central
  - CHG Cahors, Cahors, Midi Pyrennees
  - CHG St Gaudens, Saint-Gaudens, Midi Pyrennees
  - Clinique de l'Ormeau, Tarbes, Midi Pyrennees
  - CHU Purpan, Toulouse, Midi Pyrennees
  - Clinique Pasteur, Toulouse, Midi Pyrennees
  - Inst. Claudius Regaud, Toulouse, Midi Pyrennees
  - Clinique des Bonnettes, Arras, Nord
  - CH Boulogne-sur-Mer, Boulogne, Nord
  - Centre Oscar Lambret, Lille, Nord
  - Clinique des Dentellieres, Valenciennes, Nord
  - CH de Draguignan, Draguignan, Paca
  - CHI de Fréjus, Fréjus, Paca
  - Chi Frejus - St Raphael, Fréjus, Paca
  - CHICAS, Gap, Paca
  - Clinique Ste Marguerite, Hyères, Paca
  - Clinique du Cap d'Or, La Seyne-sur-Mer, Paca
  - Clinique Belvédère, Nice, Paca
  - CH Sainte Musse, Toulon, Paca
  - H.I.A Saint Anne, Toulon, Paca
  - Victor Dubos, Argenteuil, Paris Nord
  - Clinique Ste Marie, Osny, Paris Nord
  - Saint Antoine, Paris, Paris Nord
  - Saint Louis, Paris, Paris Nord
  - TENON, Paris, Paris Nord
  - Hpt Rene Dubos, Pontoise, Paris Nord
  - Clinique Porte St Cloud, Boulogne, Paris Ouest
  - BEAUJON, Clichy, Paris Ouest
  - Hopital Mignot, Le Chesnay, Paris Ouest
  - Hopital Franco Britannique, Levallois-Perret, Paris Ouest
  - Hopital Des Courses, Maisons-Laffitte, Paris Ouest
  - HARTMANN, Neuilly/seine, Paris Ouest
  - Centre Rene Huguenin, Saint-Cloud, Paris Ouest
  - Hopital Foch, Suresnes, Paris Ouest
  - Ico Angers, Angers, Pays de la Loire Region
  - Ch Cholet, Cholet, Pays de la Loire Region
  - Ch Le Mans, Le Mans, Pays de la Loire Region
  - Victor Hugo, Le Mans, Pays de la Loire Region

REFERENCES:
- [Derived] Kamioner D, Fruehauf S, Maloisel F, Cals L, Lepretre S, Berthou C. Study design: two long-term observational studies of the biosimilar filgrastim Nivestim (Hospira filgrastim) in the treatment and prevention of chemotherapy-induced neutropenia. BMC Cancer. 2013 Nov 16;13:547. doi: 10.1186/1471-2407-13-547. PMID 24237790